CLINICAL TRIAL: NCT02109848
Title: Observational Study of Keratoconus and Post-keratoplasty Eyes
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Huang, : David Huang, MD, PhD, Professor of Ophthalmology, Oregon Health and Science University, Oregon Health and Science University
Other Study IDs: OHSU IRB #00006612; R01EY018184 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-04-10 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Keratoconus and Post-keratoplasty
Keywords: keratoconus; post-keratoplasty
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- keratoconus
- post-keratoplasty
- post-DSAEK: Descemet's stripping automated endothelial keratoplasty (DSAEK)

SUMMARY:
A prospective observational study on keratoconus and post-keratoplasty will be conducted. We will enroll 50 subjects in each of 3 groups: keratoconus, post-PK, and post-DSAEK. The Optovue anterior segment OCT prototype will be used to perform 3-D corneal scans. These scans will be used to measure corneal thickness (pachymetry), corneal topography (anterior and posterior) and epithelial thickness maps. The ultrahigh-speed MIT OCT prototypes will also be used when they become available. A comprehensive eye examination, Placido-ring corneal topography, ultrasound pachymetry, and Scheimpflug camera imagery, will be performed for comparison. In some post-PK and post-DSAEK cases, vision will be primarily affected by regular astigmatism, myopia, or hyperopia, rather than HOA. These cases can be corrected by standard PRK (not OCT guided) with adjunctive mitomycin C treatment to prevent haze formation.107, 108 In these cases PRK will be performed according to the standard of care and will not be a part of the study protocol. The postoperative results will be observed at the 3-4 month visit with UCVA, manifest refraction, BSCVA, OCT scanning, Placido topography, ultrasound pachymetry, and Scheimpflug camera imagery

ELIGIBILITY:
Inclusion Criteria:

• Adults (18 & older) with keratoconus, keratoplasty, DSAEK procedures

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging.
* Inability to commit to required visits to complete the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post Operative surgical patients at Oregon Health & Science University for keratoconus, keratoplasty, DSAEK
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-06; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
validate OCT anterior topography | 3-4 month
  The primary goal of this observational study is to validate OCT anterior topography by comparison with standard Placido-ring corneal topography

CONTACTS AND LOCATIONS:
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States